CLINICAL TRIAL: NCT02828228
Title: Long-term Effects of Vitamin D Supplementation in Vitamin D Deficient Obese Children During Integrated Weight-loss Program - a Double Blind Placebo Controlled Study
Brief Title: Vitamin D Supplementation in Vitamin D Deficient Obese Children During Weight-loss Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Clinical Centre, Gdansk (Other)
Collaborators: Nutricia Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01/2016/UCK
Record Dates: First submitted 2016-06-08; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Obesity
Keywords: obesity; weight loss; vitamin D deficiency; body composition
MeSH Terms: conditions — Obesity; Weight Loss; Vitamin D Deficiency | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D 1200 IU (Experimental): Supplementation with vitamin D (1200 IU) once a day for 26 weeks
  Interventions: Drug: Vitamin D 1200 IU
- Placebo (Placebo Comparator): Placebo once a day for 26 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D 1200 IU — Vitamin D 1200 IU once a day for 26 weeks
  Other Names: cholecalciferol
  Arms: Vitamin D 1200 IU
Drug: Placebo — placebo once a day for 26 weeks
  Arms: Placebo

SUMMARY:
1. Analyze the influence of vitamin D supplementation in obese children during weight-loss program on BMI, body composition and bone mineral density.
2. Analyze the influence of vitamin D supplementation on the risk profile of obesity-related complications, namely impaired tolerance of glucose, insulin resistance, dyslipidemia and arterial hypertension, in obese children participating in weight-loss program.
3. Analyze the prevalence of vitamin D deficiency among obese children.
4. Analyze the risk factors of vitamin D deficiency in obese children (age, gender, pubertal status).

DETAILED DESCRIPTION:
The study will be conducted as a continuation and development of "6-10-14 for Health" program. The first phase of the program, financed by the municipality of Gdansk, was conducted in 2011-2013. The program comprised of screening and survey conducted among all 6-, 10- and 14-year-old children attending primary and grammar schools. A total of 18 162 children (including 7 448 6-year olds, 6 720 10-year olds and 3 994 14-year olds) were examined. A group of children with risk factors of civilization-related diseases (overweight and obesity defined according to BMI percentile charts. was identified on the basis of the screening. This group included 2 798 (16.32%) children, among them 9.17% of 6-years of age, 19.30% of 10-years and 20.48% of 14-years). All these children were qualified to intervention and education program. A total of 1 627 children qualified on the basis of screening eventually took part in the first edition of the program.

A total of 4 meetings with participating children and their caregivers were scheduled during the 12-month-long education and intervention program: at enrollment, and 3, 6 and 12 months thereafter. The meetings had form of individual consultations with various specialists. The first visit included complex medical examination, discussion on a health status of a child, interpretation of laboratory findings, and consultations with dietician, psychologist and physical education specialist. After consulting all the specialists involved in the program, individual protocol of health intervention was developed for every child. The objectives of the intervention included modification of diet, increasing health activity level and strengthening of health-seeking behaviors of child's family members. Adherence to the protocol and achieved results were evaluated during follow-up meetings with the specialists, and constituted the basis for development of individualized intervention plans for subsequent months.

The preliminary evaluation of the program effects was conducted in the group of 300 participants. The average percentile of BMI at enrollment to the program and after 12 months of participation amounted to 92.96 and 88.83, respectively. Participation in the program was reflected by a significant decrease in BMI percentile (p=0.0001), as well as by a significant drop off in fat mass content measured by bioelectrical impedance, from 39.0% to 31.4% (p=0.0001).

On the basis of these findings, the municipality of Gdansk decided to support the program for 2014-2016.

The experiment will follow a pattern of double blind randomized study. The enrolled subjects will be randomly assigned to one of the two groups:

Group 1 - weight-loss program for 52 weeks + vitamin D 1200 (IU) daily for 26 weeks Group 2 - weight-loss program for 52 weeks +placebo daily for 26 weeks

Visit I: enrollment:

* medical history, physical examination
* interpretation of laboratory findings (the tests conducted during screening + concentration of vitamin D),
* anthropometric evaluation and analysis of body composition (bioimpedance method)
* consultation of dietician, psychologist and specialist of physical activity, and defining detailed protocol of intervention
* Kasch Pulse Recovery Test
* determination of hs-C-reactive protein, Interleukin 6, chemerin and adiponectin concentrations in blood samples obtained during screening
* informing parents about the objectives and protocol of the study
* obtaining written informed consent for participation in the study
* randomization to GROUP I or II
* densitometry (DXA) - within one week after enrollment

Visit II: after 13 weeks:

* medical history, physical examination
* anthropometric evaluation and analysis of body composition (bioimpedance method)
* consultation of dietician, psychologist and specialist of physical activity, and defining detailed protocol of intervention

Within a week prior to Visit III - obtaining blood (ca. 5 ml) for laboratory testing (complete blood count, lipid profile, hs-C-reactive protein, oral glucose tolerance test, insulin, Interleukin 6, adiponectin and chemerin concentrations

Visit III: after 26 weeks:

* medical history, physical examination
* interpretation of laboratory findings
* anthropometric evaluation and analysis of body composition (bioimpedance method)
* consultation of dietician, psychologist and specialist of physical activity, and defining detailed protocol of intervention
* obtaining blood for laboratory testing
* termination of active compound/placebo administration

Visit IV: after 52 weeks:

* medical history, physical examination
* anthropometric evaluation and analysis of body composition (bioimpedance method)
* consultation of dietician, psychologist and specialist of physical activity, and defining detailed protocol of intervention
* densitometry (DXA) - within one week after terminating the study

ELIGIBILITY:
Inclusion Criteria:

* overweight (BMI between the 85th and 95th percentile) or obesity (BMI > 95th percentile), identified on the basis of anthropometric parameters
* blood concentration of 25(OH)D3 < 30 ng/ml
* written consent of legal guardians

Exclusion Criteria:

* Chronic conditions (asthma or allergies, inflammatory diseases of connective tissue, gastrointestinal disorders, diseases of kidneys and liver, disorders of bone metabolism)
* Contraindications to administration of vitamin D
* Administration of any preparation containing vitamin D, calcium, or steroid hormones during 3 months preceding the study

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 12 months
  Increase in bone mineral density during weight-loss program and vitamin D supplementation

SECONDARY OUTCOMES:
Blood level of vitamin D | 12 months
  Changes in blood level of vitamin D after supplementation
Arterial blood pressure | 12 months
  Change in blood pressure afer weight-loss and vitamin D supplementation
Lipid profile | 12 months
  Change of lipid profile after weight-loss and vitamin D supplementation
Oral Glucose Tolerance Test | 12 months
  Change of biochemical parameters after weight-loss and vitamin D supplementation
Chemerin | 12 months
  Change in chemerin level
BMI (kg/m2) | 12 months
  Change of BMI during 12-months weight loss-program and supplementation of vitamin D
Fat mass (kg) | 12 months
  Change in fat free mass during 12-months weight-loss programme and supplementation of vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Szlagatys-Sidorkiewicz, MD, PhD, Principal Investigator — University Clinical Centre, Gdansk
Locations (1):
- IUCCGdansk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Szlagatys-Sidorkiewicz A, Brzezinski M, Jankowska A, Metelska P, Slominska-Fraczek M, Socha P. Long-term effects of vitamin D supplementation in vitamin D deficient obese children participating in an integrated weight-loss programme (a double-blind placebo-controlled study) - rationale for the study design. BMC Pediatr. 2017 Apr 4;17(1):97. doi: 10.1186/s12887-017-0851-7. PMID 28376768